CLINICAL TRIAL: NCT04029025
Title: Complete Digital Workflows for the Treatment With Multiple-unit Implant-supported Fixed Dental Prostheses (iFDP): A Double-blinded Double-randomized Controlled Trial (RCT)
Brief Title: Complete Digital Workflows for the Treatment With Multiple-unit Implant-supported Fixed Dental Prostheses (iFDP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2019-00706; ex19Joda
Record Dates: First submitted 2019-07-17; First posted 2019-07-23 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Partial-edentulism; Implant-supported Fixed Dental Prostheses (iFDP)
Keywords: conventional porcelain-fused-to metal iFDP; Dentalwings DWOS Intraoral Scan; 3Shape TRIOS Pod Intraoral Scan; Dentalwings DWOS Implant Prosthetics Lab-Software; Straumann CARES Lab-Software; digital implant workflow; CAD/CAM-technology

STUDY DESIGN:
Intervention Model Description: Double-blinded double-randomized controlled trial (RCT) with crossover design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Workflow A (Active Comparator): Dentalwings DWOS Intraoral Scan (IOS A) + Dentalwings DWOS Implant Prosthetics Lab-Software (CAD A)
  Interventions: Procedure: Workflow A
- Workflow B (Active Comparator): 3Shape TRIOS Pod Intraoral Scan (IOS B) + Straumann CARES Lab-Software (CAD B)
  Interventions: Procedure: Workflow B
- Workflow C (Active Comparator): Conventional Impression + conventional porcelain-fused-to metal iFDP (LabS C/CAD C).
  Interventions: Procedure: Workflow C

INTERVENTIONS:
Procedure: Workflow A — Dentalwings DWOS Intraoral Scan (IOS A) + Dentalwings DWOS Implant Prosthetics Lab-Software (CAD A)
  Arms: Workflow A
Procedure: Workflow B — 3Shape TRIOS Pod Intraoral Scan (IOS B) + Straumann CARES Lab-Software (CAD B)
  Arms: Workflow B
Procedure: Workflow C — Conventional Impression + conventional porcelain-fused-to metal iFDP (LabS C/CAD C)
  Arms: Workflow C

SUMMARY:
This study is to assess socio-economic factors, clinical and virtual precision, patient-centered outcomes, and esthetics during the treatment with monolithic multi-unit iFDPs in a complete digital workflow

DETAILED DESCRIPTION:
Fixed Dental Prosthesis (FDPs) are the treatment of choice for the rehabilitation of partial-edentulism, especially in posterior (free-end) sites. Compared to classical tooth-bourne removable prostheses, the implant-based treatment approach is a more biological approach protecting the neighboring teeth including surrounding tissues. In addition, it is a more comfortable solution for the patient but often represents a time- and cost-intensive treatment modality.

Therefore, it is of great interest to offer the advantages of Implant-supported Fixed Dental Prosthesis (iFDP) to a broader patient population. Thus, this is only possible if new technologies are affordable, which can shorten the overall clinical treatment time and the technical production process to achieve a reasonable cost-benefit ratio in combination with a high quality outcome of the final prosthodontic reconstruction.

At this time, the classical impression technique with implant transfer posts and elastomeric materials for the manufacturing of master casts out of gypsum still represents the gold standard for implant prosthodontic reconstructions. The conventional approach involves biological, technical, patient-related and economic compromises such as complex and costly technical manufacturing steps.

An alternative to this established method is the digital implant workflow. In contrast to the conventional approach, the digital process can virtually detect the 3D implant position in a contact-free way with an Intraoral Scanner (IOS) device including further technical processing with Computer-Aided-Design (CAD)/ Computer-Aided-Manufacturing (CAM) technology.

Recently, the entire production process of monolithic iFDPs is introduced starting with IOS and following a virtual construction without any physical model situations. In addition, the production of the iFDP itself is simplified by the option to connect a full-contour monolithic Zirconium dioxide (ZrO2) reconstruction to pre-fabricated bonding base abutments in a complete digital workflow without any physical master casts.

This study is to assess socio-economic factors, clinical and virtual precision, patient-centered outcomes, and esthetics during the treatment with monolithic multi-unit iFDPs in a complete digital workflow without any physical model situation.

ELIGIBILITY:
Inclusion Criteria:

* 3-unit implant-supported Fixed Dental Prostheses (iFDP) in maxillary and mandibular sites for the replacement of premolars or molars
* at least one interproximal contact and occlusal contacts to the antagonists

Exclusion Criteria:

* uncontrolled systemic disease that would interfere with dental implant therapy
* patients who smoke > 10 cigarettes per day or tobacco equivalents
* alcohol and/or drug abuse
* patients with chronic pain
* patients with untreated periodontitis and / or inadequate oral hygiene
* medical conditions requiring chronic high dose steroid therapy or anti-resorptive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
work time (days) | from preparation to bonding of the full-contoured iFDPs to the prefabricated titanium abutments (an average of 35 days)
  work time for preparation, each production step such as computer-based design, waiting times between the various process steps, e.g. postal delivery from the external milling center, bonding of the full-contoured iFDPs to the prefabricated titanium abutments

SECONDARY OUTCOMES:
number of clinical appointments | from preparation to bonding of the full-contoured iFDPs to the prefabricated titanium abutments (an average of 35 days)
  number of clinical appointments needed for the clinical treatment steps will be recorded
chair-time in units per minutes | from preparation to bonding of the full-contoured iFDPs to the prefabricated titanium abutments (an average of 35 days)
  chair-time in units per minutes for the clinical treatment steps will be recorded
volumetric difference | at Visit 3 (an average of 30 days)
  calculation of volumetric differences for the iFDPs using the software "geomagic" (virtual accuracy measured and compared for the different workflows by means of superimposition of the gathered Standard Tessellation Language (STL)-files of each originally designed CAD-reconstruction and the secondary digitization with a laboratory scanner of all iFDPs after clinical try-in)
Change in Functional Implant Prosthodontic Score (FIPS) | at Visit 3 (an average of 30 days), Visit 4 (an average of 35 days), Visit 5 (6 months Follow-up), Visit 6 (12 months Follow-up), Visit 7 (24 months Follow-up), Visit 8 (36 months Follow-up)
  FIPS defined by 5 variables: (1) interproximal, (2) occlusion, (3) design, (4) mucosa (5) bone. Scoring scheme of 0-1-2 is assigned for each variable, resulting in a maximum score of ten (5 × 2). The variable "Interproximal" is assessed for mesial-distal contact areas and the papillary presence of the adjacent dentition. "Occlusion" is evaluated for static and dynamic patterns and "Design" for contour, shape, color and finish. The 3 variables related to restoration are scored as major discrepancy (0), minor discrepancy (1), or no discrepancy (2). Quality and quantity of peri-implant soft tissue conditions is categorized under "Mucosa" as non-keratinized/non-attached (0), non-keratinized/attached (1), or keratinized + attached (2). Marginal bone levels are analyzed under "Bone" assessing the radiographic level of the alveolar crest mesially and distally: loss > 1.5 mm (0), loss < 1.5 mm (1), and no loss (2). Higher score represents better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Joda, Prof. Dr., Principal Investigator — Universitäres Zentrum für Zahnmedizin Basel UZB, Universität Basel
Locations (1):
- Universitäres Zentrum für Zahnmedizin Basel UZB, Universität Basel, Basel, Switzerland

REFERENCES:
- [Result] Gintaute A, Weber K, Zitzmann NU, Bragger U, Ferrari M, Joda T. A Double-Blind Crossover RCT Analyzing Technical and Clinical Performance of Monolithic ZrO2 Implant Fixed Dental Prostheses (iFDP) in Three Different Digital Workflows. J Clin Med. 2021 Jun 16;10(12):2661. doi: 10.3390/jcm10122661. PMID 34208773
- [Result] Joda T, Gintaute A, Bragger U, Ferrari M, Weber K, Zitzmann NU. Time-efficiency and cost-analysis comparing three digital workflows for treatment with monolithic zirconia implant fixed dental prostheses: A double-blinded RCT. J Dent. 2021 Oct;113:103779. doi: 10.1016/j.jdent.2021.103779. Epub 2021 Aug 13. PMID 34391875